CLINICAL TRIAL: NCT06078787
Title: A Phase II Multicentric Study of Olaparib in PALB2-related Advanced Pancreatic Cancer (PALBOLA)
Brief Title: Olaparib in PALB2 Advanced Pancreatic Cancer
Acronym: PALBOLA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, CORTESI LAURA, PRINCIPAL INVESTIGATOR, Azienda Ospedaliero-Universitaria di Modena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0817L00067
Record Dates: First submitted 2023-07-06; First posted 2023-10-12 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Advanced Pancreatic Cancer; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparb (Experimental)
  Interventions: Drug: Olaparib 150 MG

INTERVENTIONS:
Drug: Olaparib 150 MG — Olaparib should be dosed 2 x 150 mg tablets (300 BID)

SUMMARY:
This is a Phase II, non-randomized, multicenter, unblinded open-label study of Olaparib in monotherapy in participants with advanced (locally advanced/metastatic) PALB2-related pancreatic cancer that have progressed after at least one treatment for advanced disease.

DETAILED DESCRIPTION:
This is a Phase II, non-randomized, multicenter, unblinded open-label study of Olaparib in monotherapy in participants with advanced (locally advanced/metastatic) PALB2-related pancreatic cancer that have progressed after at least one treatment for advanced disease.

After screening, 16 eligible participants with germline or somatic PALB2 mutations will be enrolled in this study. All participants will receive Olaparib 300 mg twice a daily (BID).

Study intervention will continue until documented PD, unacceptable AEs, intercurrent illness that prevents further administration of the study intervention, investigator's decision to discontinue the participant, participant withdrawal of consent, pregnancy of the participant, administrative reasons requiring cessation of study intervention.

After documented PD, each participant will be contacted by telephone every 12 weeks (+-14 days) to assess for survival status until withdrawal of consent to participate in the study, becoming lost to follow up, death or end of the study, whichever occurs first.

During treatment, efficacy will be evaluated using ORR, PFS, DOC and DCR using RECIST 1.1 Efficacy will also be evaluated by assessing OS. Participants will be evaluated with radiographic imaging to assess response to intervention at regular intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed pancreatic adenocarcinoma
* Has advanced (unresectable or metastatic) pancreatic cancer by American Joint Committee on Cancer 8th Edition
* Has documented mutation in PALB2 gene (germline or somatic) that is predicted to be deleterious or suspected deleterious.
* Has at least one lesion (measurable) that can be accurately assessed at baseline by CT scan (or MRI, if the subject is allergic to CT contrast media) and is suitable for repeated assessment according to RECIST Version 1.1 criteria.
* Has a life expectancy ≥16 weeks.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of either 0 or 1, as assessed within 3 days of the treatment initiation.
* Has received at least one systemic treatment for advanced disease (locally advanced or metastatic disease).
* Has adequate organ function as defined in Table 2; all screening laboratory tests should be performed within 10 days prior to initiation of study intervention.
* Is male or female, who is at least 18 years of age at the time of signing the informed consent.

Male Participants Contraceptive use by men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

* A male participant must agree to use contraception ad detailed in Appendix D of this protocol during the treatment period and for at least 3 months following the last dose of Olaparib when having sexual intercourse with pregnant woman or with a WOPBP. Female partners of male patients should also use a highly effective form of contraception ([see appendix D for acceptable methods]) if they are of childbearing potential Male patients should not donate sperm throughout the period of taking olaparib and for 3 months following the last dose of olaparib.

Female Participants Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

* 11. A female participant is eligible to participate if she is not pregnant* (Appendix D), not breastfeeding and at least 1 of the following conditions applies:

  1. Not a WOCBP as defined in Appendix D

     OR
  2. A WOCBP who agrees to follow the contraceptive guidance in Appendix D during treatment period and for least one month after the last dose of study intervention.

Postmenopausal is defined as:

* Amenorrhoeic for 1 year or more following cessation of exogenous hormonal treatments
* Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50
* radiation-induced oophorectomy with last menses >1 year ago
* chemotherapy-induced menopause with >1 year interval since last menses
* surgical sterilisation (bilateral oophorectomy or hysterectomy)

  * evidence of non-childbearing status for women of childbearing potential is defined with negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1 (within 24 hours) and before every cycles.

Informed Consent

* Has (or legally acceptable representative if applicable) provided written informed consent for the study. The participant may also provide consent/assent for future biomedical research. However, the participant may participate in the main trial without participating in the FBR.

Exclusion Criteria:

* Has a known additional malignancy that is progressing or requires active treatment. Other malignancy unless curatively treated with no evidence of disease for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
* Has myelodysplastic syndrome/acute myeloid leukaemia or features suggestive of MDS/AML.
* 3. Patients with symptomatic uncontrolled brain metastases and/or carcinomatous meningitis. Subject with previously treated brain metastasis may participate proved they are stable (without evidence of progression by imaging for at leat four weeks prior to the first dose of trial treatment and any neurological symptoms have returned to baseline), no evidence of new or enlarging brain metastases. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* 4. Has a documented weigh loss > 10% from baseline during screening and/or decline in ECOG PS to >1 between visit and within 73 hours prior to first dose of therapy.
* Has an active infection requiring systemic therapy.
* Has a known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia. Patients previously treated with Oxaliplatinum who experienced a ≤ G2 neuropathy can be included after consultation with the study physician
* Patients considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Is unable to swallow orally administered medication or patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Is a immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Has a known active hepatitis (i.e. Hepatitis B or C).

  * Active hepatitis B virus (HBV) is defined by a known positive HBV surface antigen (HBsAg) result. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.

Prior/concomitant therapy

* Any previous treatment with PARP inhibitor, including Olaparib.
* Has prior systemic chemotherapy, targeted small molecule therapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment.
* Has received prior therapy with an anti-monoclonal antibody within 4 weeks or who has not recovered (i.e. <= G1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* 15. Bone as only site of metastatic disease from pancreatic cancer (bone only disease)
* 16. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* 17. Is currently receiving known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* 18. Is currently receiving known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* 19. Has received previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* 20. Has received a whole blood transfusions in the last 120 days prior to entry to the study. Packed red blood cells and platelet transfusions are acceptable, if not performed within 28 days of the first dose of study intervention.

Prior/concurrent clinical study experience

* 21. Patients that is currently participating or has participated in another clinical study with an investigational product administered in the last 4 weeks
* 22. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.

Diagnostic assessments

* 23. Has resting ECG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* 24. Has a history or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Other exclusions

* Has a benign variant of PALB2 gene or variant of uncertain (or unknown) significance (VUS)
* Has a histology other than pancreatic adenocarcinoma (for example, neuroendocrine, adenosquamous etc.)
* Involvement in the planning and/or conduct of the study
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Is pregnant or breastfeeding,or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 30-90 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the ORR according to RECIST 1.1 following Olaparib administration | 2-3 years
  Objective response rate (ORR), defined as the percentage of patients with response of either Complete Response or Partial Response.

SECONDARY OUTCOMES:
To evaluate the PFS according to RECIST 1.1 following Olaparib administration | 2-3 years
  PFS, defined as the time from the date of the first dose until either disease progression or death due to any cause, whichever occurs first. .
To evaluate the Incidence of Treatment-Emergent Adverse Events of Olaparib | 2-3 years
  measument of Adverse events (AEs)
To evaluate the DOR according to RECIST 1.1 following Olaparib | 2-3 years
  DOR defined as the time from the date a response was first documented until either disease progression or death due to any cause, whichever occurs first.
To evaluate the DRC according to RECIST 1.1 following Olaparib | 2-3 years
  DCR defined as the percentage of patients with ORR and stable disease
To evaluate the OS according to RECIST 1.1 following Olaparib | 2-3 years
  OS definied as overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Aou Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided